CLINICAL TRIAL: NCT03869242
Title: A Prospective, Randomized, Single-center Trial of NovoTTF-200A Together With Radiation Therapy and Temozolomide Compared to Radiation Therapy and Temozolomide Alone in Patients With Newly Diagnosed GBM
Brief Title: NovoTTF-200A Together With Radiation Therapy and Temozolomide in Patients With Newly Diagnosed GBM
Acronym: NovoTTF-200A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLV-0492-18
Record Dates: First submitted 2019-02-28; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; NovoTTF-200A; Radiation Therapy; Temozolomide
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: A prospective, randomly controlled pivotal study will be conducted on 60 patients (randomized at a 1:1 ratio). Patients with histologically confirmed GBM will be randomized after debulking surgery or biopsy to either RT with concomitant TMZ and TTFields (200 kHz) for 6 weeks followed by up to 24 months of maintenance TMZ in combination with TTFields (experimental arm), or RT with concomitant TMZ alone followed by maintenance TMZ chemotherapy in combination with TTFields (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental treatment arm (Experimental): RT with concomitant TMZ and NovoTTF-200A for 6 weeks followed by up to 24 months of maintenance TMZ in combination with NovoTTF-200A.
  Interventions: Device: NovoTTF-200A
- control arm (Active Comparator): RT with concomitant TMZ alone followed by maintenance TMZ chemotherapy in combination with NovoTTF-200A.
  Interventions: Device: NovoTTF-200A

INTERVENTIONS:
Device: NovoTTF-200A — newly diagnosed GBM patients treated with NovoTTF-200A concomitant to RT and TMZ.

SUMMARY:
Study Objectives: To compare the efficacy and safety outcome of newly diagnosed GBM patients treated with NovoTTF-200A concomitant to RT and TMZ to those treated with RT and TMZ alone Study Design: Prospective, randomized, open label, standard of care control Study Hypothesis: The hypothesis of this study is that addition of NovoTTF-200A treatment to RT and TMZ will significantly increase progression free survival of newly diagnosed GBM patients compared to patients treated with RT and TMZ alone Sample Size: 60 patients with newly diagnosed GBM Study Population: Patients with tissue based diagnosis of GBM, above 18 years of age, of both genders after surgery or biopsy amenable for radiation therapy (RT) with concomitant TMZ (Stupp protocol1)

Primary endpoint:

Rate of progression-free survival at 12 months (PFS12)

Secondary endpoints:

* Overall survival (OS)
* Progression-free survival (PFS)
* Progression free survival at 6 months (PFS6)
* 1 and 2-year survival rates
* Overall radiological response (ORR, per RANO criteria)
* Safety (adverse events severity and frequency)

DETAILED DESCRIPTION:
Glioblastoma (GBM), a malignant form of astrocytoma, is the most common primary intracranial neoplasm in adults2. The incidence of GBM increases steadily above 45 years of age with a prevalence of approximately 7500 cases in the USA. Despite numerous attempts to improve the outcome of patients with GBM, the 3-year survival of patients treated with maximal surgical resection when feasible, 60 Gy radiotherapy (RT) together with concomitant temozolomide (TMZ) (RT/TMZ), followed by maintenance (adjuvant) TMZ for 6 months was only 6% with median survival of 14.6 months1. In a prospective phase 3 trial, the addition of TTFields (200 kHz) to maintenance temozolomide increased the median overall survival of patients enrolled in the study following RT/TMZ to 20.9 months, compared with 16.0 months only in the temozolomide-alone group (HR, 0.63; 95% CI, 0.53-0.76; P < .001).

TTFields are a novel treatment modality for the treatment of malignant tumors that is also referred to as the fourth modality of cancer treatment in addition to surgery, radiation therapy, and chemotherapy. Pre-clinical studies3-9 have shown this treatment modality to effectively inhibit the growth of experimental tumors both in-vitro and in-vivo without any systemic side effects. Large-scale, phase III clinical studies have validated the safety and efficacy of TTFields in patients with recurrent and newly diagnosed glioblastoma10,11. TTFields has now been approved as a standard treatment for GBM by most of the regulatory agencies around the world and its application is steadily increasing worldwide.

Standard Treatment of GBM

The currently accepted standard treatment of newly diagnosed GBM is based on: surgical resection to the extent safely feasible followed by RT with concomitant TMZ, followed by adjuvant TMZ chemotherapy in combination with TTFields. Each of these treatments is briefly described below:

1. Surgical resection - Treatment of patients with GBM usually consists of tumor resection (to the extent safely feasible) or diagnostic biopsy.
2. Radiotherapy (RT) - Post-surgical RT improves survival, though even with maximal treatment, survival after RT alone is still limited to about one year1.
3. Temozolomide (TMZ) - Concomitant TMZ chemotherapy during RT and adjuvant (maintenance) TMZ for 6 cycles has been shown to significantly improve survival (HR 0.63). This combined modality treatment is considered the standard of care.

   1. According to the TMZ (Temodar®, Temodal®) package insert adjuvant TMZ treatment delays disease progression (from 5 to 6.9 months) and improves overall survival (from 12.1 to 14.6 months)1.
   2. In the RTOG0525/EORTC Intergroup trial where patients were randomized after the end of TMZ/RT (similar to the EF-14 trial), progression-free survival was also only 6-7 months (estimated from curve)12
4. GLIADEL™ Wafers in combination with surgical resection - Gliadel™ Wafers deliver carmustine (BCNU) directly to the bed of the resected tumor. Gliadel has been approved for GBM after surgical resection, based on trials performed before TMZ therapy was established13.

   a. The package insert indicates that for newly diagnosed GBM, Gliadel™ increased median overall survival from 11.6 to 13.9 months compared to placebo. Progression-free survival with Gliadel™ wafers has been reported as 5.9 months27. No prospective data of Gliadel™ in combination with TMZ has been reported.
5. TTFields - Clinical trials of TTFields have proven safe and efficacious in patients with recurrent and newly diagnosed GBM. The median OS in the large scale phase III clinical study in newly diagnosed GBM patients (EF-14) was 20.9 months in the TTFields plus TMZ group vs. 16 months in the TMZ alone group11. Accordingly, TTFields (Optune®) are now FDA-approved for use in newly diagnosed and recurrent GBM.

In conclusion, despite the improvement in OS following the introduction of TTFields into the standard of care for newly diagnosed GBM patients, the survival of most patients remains poor. Therefore, new treatments, as well as strategies for maximizing the benefit from currently available therapies are needed.

STUDY DESIGN A prospective, randomly controlled pivotal study will be conducted on 60 patients (randomized at a 1:1 ratio). Patients with histologically confirmed GBM will be randomized after debulking surgery or biopsy to either RT with concomitant TMZ and TTFields (200 kHz) for 6 weeks followed by up to 24 months of maintenance TMZ in combination with TTFields (experimental arm), or RT with concomitant TMZ alone followed by maintenance TMZ chemotherapy in combination with TTFields (control). The primary endpoint will be rate of progression free survival at 12 months (PFS12). The sample size was chosen based on the Exact test for proportion (See XX Statistical Considerations). In short, in order to detect a PFS12 of 46.5% in patients treated with RT/TMZ/TTFields followed by maintenance TMZ+TTFields, compared to the 29.4% calculated from the EF-14 experimental arm of patients treated with RT/TMZ alone followed by maintenance TMZ+TTFields, a sample size of 60 patients randomized in a ratio of 1:1 (30 patients in each arm) is required to achieve a power of 80% at two-sided alpha level of 0.05 using the Exact test for proportion.

The following will be considered disease progression (based on the RANO criteria; Tab D):

1. 25% or more increase in enhancing lesions despite stable or increasing steroid dose
2. Increase (significant) in non-enhancing FLAIR/T2W lesions, not attributable to other non-tumor causes
3. Any new lesions Progression suspected from a clinical evaluation of the patient will need to be radiologically confirmed using an MRI scan. The criteria will not be applied in case of suspected pseudoprogression, unless the tumor continues to grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GBM according to WHO classification criteria.
* age ≥ 18 years
* Recovered from debulking surgery or biopsy-only.
* Planned treatment with RT/TMZ following maintenance TMZ (150-200 mg/m2 daily x 5 d, q28 days)
* Karnofsky performance status ≥ 70%
* Life expectancy ≥ least 3 months
* Participants of childbearing age must use effective contraception.
* All patients must sign written informed consent.
* Stable or decreasing dose of corticosteroids for the last 7 days prior to randomization, if applicable.

Exclusion Criteria:

* Early progressive disease before initiation of TMZ/RT.
* Participation in another clinical treatment trial
* Pregnancy
* Significant co-morbidities at baseline which would preclude maintenance RT or TMZ treatment, as determined by the investigator:
* Thrombocytopenia (platelet count < 100 x 103/μL)
* Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
* CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
* Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
* Total bilirubin > 1.5 x upper limit of normal
* Significant renal impairment (serum creatinine > 1.7 mg/dL, or > 150 µmol/l)
* Implanted pacemaker, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* History of hypersensitivity reaction to TMZ or a history of hypersensitivity to DTIC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS12 | 12 months
  Rate of progression-free survival at 12 months

SECONDARY OUTCOMES:
PFS6 | 6 months
  Progression-free survival at 6 months
One and two year survival rate | 24 months
  One and two year survival rate
Radiological response | 24 months
  ORR- Overall Radiological response.
adverse events | 36 months
  adverse events severity and frequency
Radiological response | 26 months
  RANO - response assessment in neuro-oncology

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv saurasky medical center, Tel Aviv, Israel